CLINICAL TRIAL: NCT00599105
Title: Angiogenesis in Early Breast Cancer for Prognosis Prediction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Min-Ying Su, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCI-HS-2000-1141; NIH-CA90437; CBCRP-9WB-0020
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Breast Lesions
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: magnetic resonance imaging — MRI contrast agent, 0.1 mmol/kg

SUMMARY:
This study will investigate the association of angiogenesis in breast cancer measured by magnetic resonance imaging and biomarkers with long-term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a breast mass highly suspicious for malignancy from clinical, mammographic or sonographic examination.
* The study has been explained to the patient when she is scheduled for surgery.
* Healthy normal volunteers for imaging protocol optimization.

Exclusion Criteria:

* Pregnancy
* Patients with implanted surgical clips (hemostatic clips) or other ferromagnetic material,
* Patients engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials, or who may have imbedded metal fragments from military activities,
* Patients with metallic implants, because they may cause artifacts in diagnostic images due to magnetic field distortion,
* Patients with implanted prosthetic heart valves,
* Patients with pacemakers, neuro-stimulation devices,
* A breast mass with features of benign tumor
* The patients unwilling to participate in the study or fail to sign the consent form

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2000-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To investigate whether breast cancer with a higher angiogenesis activity is associated with a unfavorable outcome. | 5 years from completion of enrollment

SECONDARY OUTCOMES:
To investigate whether angiogenesis of breast cancer is associated wit lymph node status | at completion of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Functional Onco-Imaging, University of California, Irvine, California, United States